CLINICAL TRIAL: NCT01956266
Title: Treatment of Emotional Prosodic Disorders in Parkinson's Disease
Brief Title: Emotional Prosody Treatment in Parkinson's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O0958-M
Record Dates: First submitted 2013-09-13; First posted 2013-10-08 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease
Keywords: Prosody; Communication; Dysarthria
MeSH Terms: conditions — Parkinson Disease; Communication; Dysarthria

STUDY DESIGN:
Intervention Model Description: Single group, pretest postest behavioral treatment design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Emotional prosodic treatment (Experimental): The experimental treatment is consistent with the standard treatment in that it targets impairments in pitch/stress, loudness variability and control of speech rate, the core characteristics of prosodic insufficiency in PD (Darley, Aronson & Brown, 1969). However, the experimental treatment provides an innovative and targeted emphasis on the emotional component of the disorder. The production of emotional intonation in an utterance requires varying combinations of pitch/stress, loudness, and rate.
  Interventions: Behavioral: Emotional prosodic treatment

INTERVENTIONS:
Behavioral: Emotional prosodic treatment — The experimental treatment is consistent with the standard treatment in that it targets impairments in pitch/stress, loudness variability and control of speech rate, the core characteristics of prosodic insufficiency in PD (Darley, Aronson & Brown, 1969). However, the experimental treatment provides an innovative and targeted emphasis on the emotional component of the disorder. The production of emotional intonation in an utterance requires varying combinations of pitch/stress, loudness, and rate. Participants will receive clinician feedback as well as auditory and visual feedback on accuracy via the VisiPitch display.

SUMMARY:
This study investigates a treatment protocol which holds the potential to significantly improve communication and quality of life for individuals affected by Parkinson's disease (PD). Disorders of emotional communication are widely reported in PD and can negatively impact quality of life by increasing social isolation and decreasing independence. Individuals with emotional prosodic communication disorders are often perceived as depressed or unconcerned about others. This seeming negativity can cause difficulties in relationships, and increased feelings of stress and burden in caregivers which may result in earlier placement in an institutional care setting. This innovative treatment program could improve care for individuals with PD, as well as other individuals who may be affected by disorders of emotional prosodic communication (e.g., stroke or traumatic brain injury).

DETAILED DESCRIPTION:
Individuals with Parkinson's disease (PD) present with a variety of motor symptoms including resting tremor, difficulty initiating movement/slowed movements, and rigidity. While these motor signs and symptoms are the hallmark features, individuals with PD also often demonstrate changes in communication ability, with an estimated prevalence of 89 percent of all individuals with PD being affected. These disorders of communication have been reported by individuals with PD and their caregivers to be one of the most difficult aspects of living with this disorder.

The most commonly diagnosed communicative disorder in PD is hypokinetic dysarthria which can result in changes in prosody, respiratory control, voice quality, and articulation. Of these, the disorders in prosody have been judged to be the most prominent deficit. Prosody includes the pitch, loudness, and rate with which speech utterances are produced and is used to communicate emotional connotation (e.g. angry versus sad). Impairments in speech prosody reduce the ability to communicate emotional feelings or intentions as well as reducing the intelligibility of the spoken message. While pharmacological treatments have been shown to be effective in improving motor function, these medications have not been shown to greatly mitigate speech production disorders including prosody, suggesting that therapies other than dopaminergic agents are needed to address prosody deficits in PD. Despite a negative impact on quality of life and reduced independence of individuals affected by emotional prosodic disorders, no published studies are available testing therapies to improve production of emotional prosody in PD.

The primary goal of this proposal is to compare a treatment protocol shown to be effective in treating emotional prosodic deficit in stroke and TBI (Leon et al., 2005; Rosenbek et al., 2006) to a standard clinical treatment for prosody deficit that does not target the emotional aspect of the disorder in individuals with PD. The experimental treatment targets increased pitch and loudness variability, and control of speech rate, the core characteristics of prosodic insufficiency in PD, but with an emphasis on the emotional component of the disorder. The primary aims of the study are to determine treatment effect size by measuring the difference of the experimental protocol versus standard clinical care on prosodic deficit in individuals with PD via changes in acoustic and perceptual measures, as well as provide psychometric validation of test-retest reliability of the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Experimental subjects must meet the Brain Bank criteria (Gibb & Lees, 1988) for idiopathic PD.
* All participants must:

  * be between the ages of 45 and 85
  * have at least a sixth grade education
  * fluent in English
* The investigators will obtain information about participant's Parkinson's disease history from medical records including:

  * age at onset
  * current age
  * gender
  * handedness
  * level of education
  * side of the body initially affected
  * information regarding subsequent clinical progression
  * medications
  * most recent Unified Parkinson Disease Rating Scale (UPDRS) scores
  * Hoehn and Yahr (H&Y) (Hoehn & Yahr, 1967) scores
* The investigators will include subjects with H&Y Stages between 2 and 4
* Participants must be judged as having at least a mild level of affective prosodic deficit in pretreatment testing

Exclusion Criteria:

* Individuals will be excluded with other forms of Parkinsonism such as:

  * multiple systems atrophy
  * Lewy body dementia
  * progressive supranuclear palsy
* Other exclusionary criteria will be:

  * co-existing dementia (as indicated by score on Montreal Cognitive Assessment of below 26)
  * neurological disease other than idiopathic PD
  * major depression
  * any other psychiatric illness
  * chronic medical and neurological diseases other than PD (e.g., cardiac failure, renal disease, hepatic failure, stroke, or severe sensory deficits such as deafness or blindness (corrected visual acuity less than 20/50).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change from pre to post treatment in perceptual and acoustic analysis of sentences spoken in emotional tones. | Administered before initiation of treatment and after 8 treatment sessions over an expected average of 3 weeks.
  The primary outcome of 96 semantically neutral sentences is read aloud using one of four emotional tones of voice. The participant will be given a card with the sentence and a card denoting the emotional tone to be used when speaking the sentence aloud. Participants will be wearing a headset cardioid microphone with frequency response tailored to vocal use with a shock mount to reduce handling and cable noise. Participant's responses will be recorded using the VisiPitch IV software designed for analysis and feedback and stored for future analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Leon, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-08-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT01956266/SAP_000.pdf
  • Informed Consent Form (2014-06-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT01956266/ICF_001.pdf